CLINICAL TRIAL: NCT00281749
Title: Telephone Call From Acute Care Physicians to Long Term Care Physicians: Impact on Transitional Care of Elderly Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05/12/VA03
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Alzheimer Disease; Parkinson Disease; Dysphagia
Keywords: ALZHEIMER'S D-SE; PARKINSON'S D-SE; FRAILTY
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Deglutition Disorders; Frailty

INTERVENTIONS:
Procedure: TELEPHONE CALL

SUMMARY:
A telephone call from a physician taking care of a patient in the hospital to a physician in the long term care setting at the time of discharge can improve transitional care for elderly patients. We believe direct communication between physicians can reduce re-hospitalizations, medication errors, morbidity and mortality. No studies have been done that involve physician-to-physician sign-outs after hospital discharge to the nursing home. In our study, we would like to address the breakdown in the transfer of information to the nursing home setting.

ELIGIBILITY:
Inclusion Criteria:

* patients transitioning from the Acute Care for The Elderly (ACE) Unit patients at Maimonides Medical Center to Metropolitan Jewish Geriatric Center (MJGC).

Exclusion Criteria:

* AGE BELOW 65

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SERGEY I GENKIN, MD, Principal Investigator — Maimonides Medical Center
Locations (2):
- United States (2):
  - Maimonide Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York